CLINICAL TRIAL: NCT00125450
Title: Efficacy and Safety of Chest Physiotherapy With Forced Expiratory Technique for Acute Bronchiolitis in Toddlers
Brief Title: Evaluation of Chest Physiotherapy for Acute Bronchiolitis in Toddlers (BRONKINOU)
Acronym: BRONKINOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association des Réseaux Bronchiolite (Unknown)
Responsible Party: Marc LEGRAND, Department Clinical Research of Developpemnt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P030421; AOM 03123; DGS 2004/0276
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2006-10

CONDITIONS: Viral Bronchiolitis
Keywords: Acute Bronchiolitis; Chest Physiotherapy; Forced Expiratory Techniques; Double Blind Trial; Children; Pediatric; RESPIRATORY SYNCYTIAL VIRUS
MeSH Terms: conditions — Bronchiolitis, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Chest Physiotherapy with Forced Expiratory Technique
  Interventions: Procedure: Chest Physiotherapy with Forced Expiratory Technique
- B (Active Comparator): Aspiration
  Interventions: Procedure: Nasopharyngeal Aspiration

INTERVENTIONS:
Procedure: Chest Physiotherapy with Forced Expiratory Technique — Chest Physiotherapy with Forced Expiratory Technique
  Other Names: A. Chest Physiotherapy with Forced Expiratory Technique
  Arms: A
Procedure: Nasopharyngeal Aspiration — Nasopharyngeal Aspiration
  Arms: B

SUMMARY:
The purpose of this study is to determine whether chest physiotherapy with forced expiratory technique reduces delay of healing in acute bronchiolitis of children between 15 days and 24 months of age.

DETAILED DESCRIPTION:
Bronchiolitis is the most common lower respiratory infection in infants, and the respiratory condition leading to the majority of hospital admissions in young children. It is also probably the most common serious illness of childhood lacking evidence-based treatment. Evidence against the effectiveness of chest physiotherapy with vibration and postural drainage techniques has been described but forced expiratory technique, as described in France, has never been evaluated.

The investigators hypothesised that forced expiratory technique was able to reduce the duration of respiratory distress.

Comparison(s): The investigators compare physiotherapy with forced expiratory techniques to simple aspiration of naso-pharyngeal secretions.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 15 days to 24 months
* First acute bronchiolitis
* Indication of hospitalisation
* One or more of these criteria : toxic aspect; apnea or cyanosis; respiratory rate > 60/min; pulse oxymetry < 95%; alimentary intake < 2/3 of the needs.

Exclusion Criteria:

* Prematurity (gestational age < 32 weeks)
* Brondysplasia
* Chronic lung disease or congenital heart disease
* Respiratory distress necessitating admission in the Pediatric Intensive Care Unit (PICU)
* 3 or more chest physiotherapy procedures since hospitalisation
* Parental refusal
* Any chest physiotherapy contra-indication

Ages: 15 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2004-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Delay for obtention of healing defined by all of these parameters at least 8 hours in a row : pulse oxymétry >94% AND normal feeding AND specific respiratory distress score lower than one as described in the protocol AND normal respiratory rate | obtention

SECONDARY OUTCOMES:
Safety of the forced expiratory technique | during hospitalisation
Comparison of pulse oxymetry before/after chest physiotherapy | during hospitalisation
Quality of Life Scale | on discharge

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gajdos, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Philippe Labrune, MD - PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (7):
- France (7):
  - Jean Verdier Hospital, Bondy
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Antoine Béclère Hospital - Pediatric Department, Clamart
  - Kremlin Bicetre Hospital, Le Kremlin-Bicêtre
  - Trousseau Hospital, Paris
  - Necker - Enfants Malades Hospital, Paris
  - Robert Debré Hospital, Paris

REFERENCES:
- [Background] Perrotta C, Ortiz Z, Roque M. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD004873. doi: 10.1002/14651858.CD004873.pub2. PMID 15846736
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196
- [Derived] Gajdos V, Katsahian S, Beydon N, Abadie V, de Pontual L, Larrar S, Epaud R, Chevallier B, Bailleux S, Mollet-Boudjemline A, Bouyer J, Chevret S, Labrune P. Effectiveness of chest physiotherapy in infants hospitalized with acute bronchiolitis: a multicenter, randomized, controlled trial. PLoS Med. 2010 Sep 28;7(9):e1000345. doi: 10.1371/journal.pmed.1000345. PMID 20927359
- See also: sponsor web site — http://www.aphp.fr